CLINICAL TRIAL: NCT06444425
Title: Korotkoff Sounds Dynamically Reflect Changes in Cardiac Function Based on Deep Learning Methods: A Prospective, Multicenter Study
Brief Title: Artificial Intelligence in Detecting Cardiac Function
Status: Enrolling by invitation | Type: Observational
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Collaborators: Zhejiang Taizhou hospital (Unknown); The People's Hospital of Quzhou (Other); Zhejiang Quhua Hospital (Other); Hong Kong Applied Science and Technology Research Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: KY-2024-108
Record Dates: First submitted 2024-05-31; First posted 2024-06-05 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure; Deep Learning
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heart Failure: Patients with stable heart failure were defined as those with structural heart disease and a history of heart failure episodes but no current symptoms or signs of heart failure after receiving anti-heart failure treatment during hospitalization, such as decreased exercise tolerance (dyspnea, fatigue), fluid retention, etc. Additionally, according to the 2024 Chinese guidelines for the diagnosis and treatment of heart failure consensus, patients eligible for this study will be classified based on ejection fraction into the following categories:
  * Reduced ejection fraction heart failure (HFrEF): HFrEF is defined by LVEF < 40%
  * Preserved ejection fraction heart failure (HFpEF): HFpEF is defined by LVEF ≥ 50%
  * Heart failure with mid-range ejection fraction (HFmrEF): HFmrEF refers to heart failure characterized by LVEF between 40% and 49%.
- Normal: There were no structural or functional abnormalities in the cardiac system, and no symptoms or signs of heart failure were observed. Alternatively, the patient has developed organic heart disease without exhibiting any symptoms or signs of heart failure.

SUMMARY:
The Korotkoff Sounds（KS）, which have been in use for over a century, are widely regarded as the gold standard for measuring blood pressure. Furthermore, their potential extends beyond diagnosis and treatment of cardiovascular disease; however, research on the KS remains limited. Given the increasing incidence of heart failure (HF), there is a pressing need for a rapid and convenient prehospital screening method. In this study, we propose employing deep learning (DL) techniques to explore the feasibility of utilizing KS methodology in predicting functional changes in cardiac ejection fraction (LVEF) as an indicator of cardiac dysfunction.

DETAILED DESCRIPTION:
Blood Pressure Measurement：Around 72 hours before and after the completion of the patient's echocardiogram, considering the variability in the patient's blood pressure and ejection fraction at different times, blood pressure should be measured in each participant at least twice a day, up to a maximum of six times. Each patient should be instructed to remain in a quiet state for 10 minutes before blood pressure measurement. Blood pressure measurement should be conducted according to the following criteria: the cuff used to measure blood pressure should be wrapped around the patient's arm above the elbow joint, positioned 2-3 cm above the level of the heart, with a snugness that allows one finger to fit underneath. Place the stethoscope head at the brachial artery pulse point on the left elbow joint, then begin inflation. Inflate continuously until the sound of the pulse beat disappears; then inflate an additional 20 mmHg before stopping inflation. Slowly deflate while listening-the first audible pulse beat is the systolic pressure, and the disappearance of the pulse sound is the diastolic pressure. Use the Hanhong POPULAR-3 electronic stethoscope to record the aforementioned process, with each audio recording lasting 25 seconds uniformly.

Data Analysis Overview:

In terms of data analysis, deep learning models are developed based on Torch version 1.5.0, utilizing Transformer network architecture to analyze the collected audio data.

Network One: Identifying the presence of cardiac functional abnormalities through Korotkoff sounds.

Evaluation Metrics: Receiver Operating Characteristic (AUROC), sensitivity, specificity, and F1 score (harmonic mean of sensitivity and specificity) to assess model performance on the test dataset.

Network Two: NYHA classification of Korotkoff sounds. Evaluation Metrics: Confusion matrix, weighted accuracy, multi-class ROC curve, F1 score.

Network Three: Heart failure classification of Korotkoff sounds in heart failure patients.

Evaluation Metrics: Confusion matrix, weighted accuracy, multi-class ROC curve, F1 score.

Network Four: Left Ventricular Ejection Fraction (LVEF) prediction from Korotkoff sounds.

Evaluation Metrics: Root Mean Squared Error (RMSE), Mean Absolute Error (MAE), Mean Squared Error (MSE), R2 Score.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were admitted to the Cardiology Department of the aforementioned four Groups (The Fourth Affiliated Hospital of School of Medicine of Zhejiang University, Zhejiang Taizhou Hospital, Quzhou People's Hospital, Zhejiang Quhua Hospital)between June 2024 and December 2024, and successfully underwent echocardiographic examinations.
2. Individuals aged between 18 and 90 years with a resting heart rate ranging from 60 to 100 beats per minute.
3. Demonstrating good compliance, capable of cooperating in completing multiple blood pressure measurements within 72 hours following the completion of echocardiography.
4. Willingness to voluntarily participate in the study.

Exclusion Criteria:

1. Patients with acute decompensated heart failure, acute myocardial infarction, atrioventricular block;
2. Cerebral hemorrhage, severe infection, active digestive tract ulcer, severe hematological diseases, severe liver and kidney dysfunction or other serious medical or surgical conditions;
3. Pregnant or lactating women;
4. Patients with mental illness;
5. Individuals who have participated in other clinical trials within the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were admitted to the Cardiology Department of the aforementioned four Groups (The Fourth Affiliated Hospital of School of Medicine of Zhejiang University, Zhejiang Taizhou Hospital, Quzhou People's Hospital, Zhejiang Quhua Hospital) between June 2024 and December 2024, and successfully underwent echocardiographic examinations.
Sampling Method: Probability Sample
Enrollment: 685 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac Dysfunction | Evaluation LVEF：Cardiac ultrasound was performed 72 hours prior to and following anti-Acute Heart Failure treatment.
  The pathophysiology of heart failure encompasses a multifaceted clinical syndrome: 1)Cardiac structural and/or functional abnormalities resulting in impaired ventricular diastolic function and/or systolic ejection capacity;2)Corresponding clinical manifestations indicative of heart failure; 3)Typically accompanied by elevated levels of beneficial natriuretic peptide(BNP), as well as pulmonary or systemic congestion suggestive of cardiac origin on imaging studies, or objective evidence of increased ventricular filling pressure on hemodynamic assessments.4)According to the classification of left ventricular ejection fraction (LVEF) based on cardiac ultrasound, heart failure can be categorized into four types: reduced ejection fraction heart failure (HFrEF), improving ejection fraction heart failure (HFimpEF), moderately reduced ejection fraction heart failure (HFmrEF), and retained ejection fraction heart failure (HFpEF).

CONTACTS AND LOCATIONS:
Overall Officials: Sixiang Jia, MD, Study Director — The fourth hospital affiliated to zhejiang university school of medicine
Locations (1):
- The Fourth Hospital Affiliated to Zhejiang University School of Medicine, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No